CLINICAL TRIAL: NCT03217565
Title: A Phase 1, Single- and Multiple-Dose Safety and Pharmacokinetic Study of Oral and IV Tedizolid Phosphate (MK-1986) in Inpatients Under 2 Years Old
Brief Title: A Pharmacokinetic Study of Tedizolid Phosphate in Pediatric Participants With Gram-Positive Infections (MK-1986-014)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1986-014; MK-1986-014 (Other: MSD Protocol Number); 2017-000953-38 (EudraCT Number)
Record Dates: First submitted 2017-07-12; First posted 2017-07-14 (Actual); Results first posted 2024-07-22 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-01

CONDITIONS: Gram-Positive Infections
MeSH Terms: interventions — tedizolid phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Part A Group 1 Cohort 1: Single Dose IV Tedizolid Phosphate 28 days to <6 months (Experimental): Pediatric participants 28 days to <6 months of age will receive a single dose (SD) intravenous (IV) infusion of tedizolid phosphate according to body weight: 3 mg/kg for body weight <10 kg or 2.5 mg/kg for body weight 10 to <30 kg.
  Interventions: Drug: IV Tedizolid Phosphate
- Part A Group 1 Cohort 2: Single Dose IV Tedizolid Phosphate 6 months to <24 months (Experimental): Pediatric participants 6 months to <24 months of age will receive an SD IV infusion of tedizolid phosphate according to body weight: 3 mg/kg for body weight <10 kg or 2.5 mg/kg for body weight 10 to <30 kg.
  Interventions: Drug: IV Tedizolid Phosphate
- Part A Group 2 Cohort 1: Single Dose IV Tedizolid Phosphate (full term) birth to <28 days (Experimental): Full term (FT) neonates from birth to <28 days of age will receive an SD IV infusion of tedizolid phosphate according to body weight: 3 mg/kg for body weight <10 kg or 2.5 mg/kg for body weight 10 to <30 kg.
  Interventions: Drug: IV Tedizolid Phosphate
- Part A Group 2 Cohort 2: Multiple Dose IV Tedizolid Phosphate (full term) birth to <28 days (Experimental): FT neonates from birth to <28 days of age will receive multiple dose (MD) IV infusions of tedizolid phosphate according to body weight: 3 mg/kg for body weight <10 kg or 2.5 mg/kg for body weight 10 to <30 kg, administered twice daily for 3 days.
  Interventions: Drug: IV Tedizolid Phosphate
- Part A Group 3 Cohort 1: Single Dose IV Tedizolid Phosphate (preterm) birth to <28 days (Experimental): Preterm (PT) neonates from birth to <28 days of age will receive an SD IV infusion of tedizolid phosphate according to body weight: 3 mg/kg for body weight <10 kg or 2.5 mg/kg for body weight 10 to <30 kg.
  Interventions: Drug: IV Tedizolid Phosphate
- Part A Group 3 Cohort 2: Multiple Dose IV Tedizolid Phosphate IV (preterm) birth to <28 days (Experimental): PT neonates from birth to <28 days of age will receive MD IV infusions of tedizolid phosphate according to body weight: 3 mg/kg for body weight <10 kg or 2.5 mg/kg for body weight 10 to <30 kg, administered twice daily for 3 days.
  Interventions: Drug: IV Tedizolid Phosphate
- Part B Group 4: Single Dose Oral Tedizolid Phosphate 28 days to <24 months (Experimental): Pediatric participants 28 days to <24 months of age will receive an SD oral suspension of tedizolid phosphate according to body weight: 3 mg/kg for body weight <10 kg or 2.5 mg/kg for body weight 10 to <30 kg.
  Interventions: Drug: Oral Suspension Tedizolid Phosphate
- Part B Group 5: Single Dose Oral Tedizolid Phosphate (full term) birth to <28 days (Experimental): FT neonates from birth to <28 days of age will receive an SD oral suspension of tedizolid phosphate according to body weight: 3 mg/kg for body weight <10 kg or 2.5 mg/kg for body weight 10 to <30 kg.
  Interventions: Drug: Oral Suspension Tedizolid Phosphate
- Part B Group 6: Single Dose Oral Tedizolid Phosphate (preterm) birth to <28 days (Experimental): PT neonates from birth to <28 days of age will receive an SD oral suspension of tedizolid phosphate according to body weight: 3 mg/kg for body weight <10 kg or 2.5 mg/kg for body weight 10 to <30 kg.
  Interventions: Drug: Oral Suspension Tedizolid Phosphate

INTERVENTIONS:
Drug: IV Tedizolid Phosphate — A single dose, or twice daily dose for 3 days, of tedizolid phosphate administered IV.
  Arms: Part A Group 1 Cohort 1: Single Dose IV Tedizolid Phosphate 28 days to <6 months; Part A Group 1 Cohort 2: Single Dose IV Tedizolid Phosphate 6 months to <24 months; Part A Group 2 Cohort 1: Single Dose IV Tedizolid Phosphate (full term) birth to <28 days; Part A Group 2 Cohort 2: Multiple Dose IV Tedizolid Phosphate (full term) birth to <28 days; Part A Group 3 Cohort 1: Single Dose IV Tedizolid Phosphate (preterm) birth to <28 days; Part A Group 3 Cohort 2: Multiple Dose IV Tedizolid Phosphate IV (preterm) birth to <28 days
Drug: Oral Suspension Tedizolid Phosphate — A single dose of tedizolid phosphate administered as an oral suspension.
  Arms: Part B Group 4: Single Dose Oral Tedizolid Phosphate 28 days to <24 months; Part B Group 5: Single Dose Oral Tedizolid Phosphate (full term) birth to <28 days; Part B Group 6: Single Dose Oral Tedizolid Phosphate (preterm) birth to <28 days

SUMMARY:
The primary objectives of this study are to describe the single-dose, and multiple dose pharmacokinetics (PK) of intravenous (IV) tedizolid phosphate, or a single dose oral suspension of tedizolid phosphate, when administered to pediatric participants, full-term neonates, and preterm neonates.

DETAILED DESCRIPTION:
Per protocol, PK analysis in Part A Group 1 will be conducted across ages in Cohorts 1 and 2 combined: Part A Group 1 Cohort 1 + Cohort 2: 28 days to <24 months.

ELIGIBILITY:
Inclusion Criteria:

* Is receiving prophylaxis for or has a confirmed or suspected infection with gram-positive bacteria and receiving concurrent antibiotic treatment with gram -positive antibacterial activity.
* Is at least 1 kg in weight.
* Is in stable condition as determined from medical history, physical examination, electrocardiogram (ECG), vital signs, and clinical laboratory evaluations.
* Has no clinically significant ECG abnormalities.
* Has sufficient vascular access to receive trial drug, and allow for required blood draws.
* Is able to receive medication by mouth, for those dosed with oral suspension; dose administration via feeding tube is acceptable.

Exclusion Criteria:

* Has a history of seizures, other than febrile seizures, clinically significant cardiac arrhythmia or condition, moderate or severe renal impairment, or any physical condition that could interfere with the interpretation of the study results, as determined by the Investigator.
* Has used rifampin within 14 days prior to dosing.
* Has used or will be using proton pump inhibitors, H2 blockers, or antacids (for participants in Part B, i.e, oral suspension dose) at any time from 24 hours prior to dosing through 24 hours after dosing..
* Has a recent (3-month) history or current infection with viral hepatitis or other significant hepatic disease.
* Has a history of drug allergy or hypersensitivity to oxazolidinones.
* Has had significant blood loss.
* Need for oral administration of topotecan, rosuvastatin, irinotecan, or methotrexate during administration of oral study drug.
* Used monoamine oxidase inhibitors (MAOIs) or serotonergic agents including tricyclic antidepressants, selective serotonin reuptake inhibitors (SSRIs), and serotonin 5-hydroxytryptamine receptor agonists (triptans), meperidine, or buspirone within 14 days prior to study, or planned use while on study.
* Has received another investigational product within the 30 days prior to enrollment.

Ages: 1 Day to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2023-03-18 (Actual); Study Completion 2023-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (30):
- United States (7):
  - Arkansas Children's Hospital ( Site 1012), Little Rock, Arkansas
  - Children's Hospital of Orange County ( Site 1001), Orange, California
  - Sharp Memorial Hospital ( Site 1021), San Diego, California
  - Ann & Robert H. Lurie Children's Hospital of Chicago ( Site 1022), Chicago, Illinois
  - Our Lady of the Lake Regional Medical Center. ( Site 1004), Baton Rouge, Louisiana
  - Saint Louis Children's Hospital ( Site 1020), St Louis, Missouri
  - Primary Children's Hospital ( Site 1000), Salt Lake City, Utah
- Bulgaria (11):
  - Medical Center - 1- Sevlievo EOOD ( Site 2207), Sevlievo, Gabrovo
  - MHAT Sv. Ivan Rilski EOOD ( Site 2201), Kozloduy, Vratsa
  - UMHAT Deva Maria ( Site 2208), Burgas
  - MHAT Dr. Tota Venkova-Pediatrics ( Site 2218), Gabrovo
  - MHAT "Dr. Stamen Iliev" Montana ( Site 2215), Montana
  - MHAT City Clinic Sv. Georgi EOOD ( Site 2202), Montana
  - UMHAT Dr. Georgi Stranski EAD ( Site 2211), Pleven
  - MHAT Rousse-Neonatology ( Site 2213), Rousse
  - Multiprofile Hospital for Active Treatment - Ruse ( Site 2204), Rousse
  - UMHAT Kanev AD ( Site 2209), Rousse
  - MHAT Dr. Ival Seliminski ( Site 2212), Sliven
- Colombia (4):
  - Hospital San Vicente Fundacion ( Site 1103), Medellín, Antioquia
  - Clinica de la Costa S.A.S. ( Site 1106), Barranquilla, Atlántico
  - Fundacion Hospital Infantil Universitario de San Jose ( Site 1107), Bogotá, Bogota D.C.
  - Fundacion Valle del Lili ( Site 1102), Cali, Valle del Cauca Department
- Norway (4):
  - Akershus Universitetssykehus HF ( Site 1604), Loerenskog, Akershus
  - Haukeland Universitetssjukehus ( Site 1602), Bergen, Hordaland
  - Stavanger Universitetssykehus, Helse Stavanger ( Site 1601), Stavanger, Rogaland
  - St. Olavs Hospital. ( Site 1600), Trondheim, Sor-Trondelag
- United Kingdom (4):
  - University Hospital Southampton NHS Foundation Trust ( Site 1700), Southampton, Hampshire
  - Alder Hey Childrens NHS Foundation Trust Hospital ( Site 1703), Liverpool, Lancashire
  - Royal Victoria Infirmary ( Site 1702), Newcastle, Newcastle Upon Tyne
  - Oxford University Hospitals NHS Foundation Trust ( Site 1704), Oxford, Oxfordshire

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 30 centers in 5 countries.
Groups:
- Part A Group 1 Cohort 1: Single Dose IV Tedizolid Phosphate 28 Days to <6 Months: Pediatric participants 28 days to <6 months of age received a single dose (SD) intravenous (IV) infusion of tedizolid phosphate according to body weight: 3 mg/kg for body weight <10 kg or 2.5 mg/kg for body weight 10 to <30 kg.
- Part A Group 1 Cohort 2: Single Dose IV Tedizolid Phosphate 6 Months to <24 Months: Pediatric participants 6 months to <24 months of age received an SD IV infusion of tedizolid phosphate according to body weight: 3 mg/kg for body weight <10 kg or 2.5 mg/kg for body weight 10 to <30 kg.
- Part A Group 2 Cohort 1: Single Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days: Full term (FT) neonates from birth to <28 days of age received an SD IV infusion of tedizolid phosphate according to body weight: 3 mg/kg for body weight <10 kg or 2.5 mg/kg for body weight 10 to <30 kg.
- Part A Group 2 Cohort 2: Multiple Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days: FT neonates from birth to <28 days of age received multiple dose (MD) IV infusions of tedizolid phosphate according to body weight: 3 mg/kg for body weight <10 kg or 2.5 mg/kg for body weight 10 to <30 kg, administered twice daily for 3 days.
- Part A Group 3 Cohort 1: Single Dose IV Tedizolid Phosphate (Preterm) Birth to <28 Days: Preterm (PT) neonates from birth to <28 days of age received an SD IV infusion of tedizolid phosphate according to body weight: 3 mg/kg for body weight <10 kg or 2.5 mg/kg for body weight 10 to <30 kg.
- Part A Group 3 Cohort 2: Multiple Dose IV Tedizolid Phosphate IV (Preterm) Birth to <28 Days: PT neonates from birth to <28 days of age received MD IV infusions of tedizolid phosphate according to body weight: 3 mg/kg for body weight <10 kg or 2.5 mg/kg for body weight 10 to <30 kg, administered twice daily for 3 days.
- Part B Group 4: Single Dose Oral Tedizolid Phosphate 28 Days to <24 Months: Pediatric participants 28 days to <24 months of age received an SD oral suspension of tedizolid phosphate according to body weight: 3 mg/kg for body weight <10 kg or 2.5 mg/kg for body weight 10 to <30 kg.
- Part B Group 5: Single Dose Oral Tedizolid Phosphate (Full Term) Birth to <28 Days: FT neonates from birth to <28 days of age received an SD oral suspension of tedizolid phosphate according to body weight: 3 mg/kg for body weight <10 kg or 2.5 mg/kg for body weight 10 to <30 kg.
- Part B Group 6: Single Dose Oral Tedizolid Phosphate (Preterm) Birth to <28 Days: PT neonates from birth to <28 days of age received an SD oral suspension of tedizolid phosphate according to body weight: 3 mg/kg for body weight <10 kg or 2.5 mg/kg for body weight 10 to <30 kg.
Period: Overall Study
Arm/Group | Part A Group 1 Cohort 1: Single Dose IV Tedizolid Phosphate 28 Days to <6 Months | Part A Group 1 Cohort 2: Single Dose IV Tedizolid Phosphate 6 Months to <24 Months | Part A Group 2 Cohort 1: Single Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 2 Cohort 2: Multiple Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 3 Cohort 1: Single Dose IV Tedizolid Phosphate (Preterm) Birth to <28 Days | Part A Group 3 Cohort 2: Multiple Dose IV Tedizolid Phosphate IV (Preterm) Birth to <28 Days | Part B Group 4: Single Dose Oral Tedizolid Phosphate 28 Days to <24 Months | Part B Group 5: Single Dose Oral Tedizolid Phosphate (Full Term) Birth to <28 Days | Part B Group 6: Single Dose Oral Tedizolid Phosphate (Preterm) Birth to <28 Days
Started | 4 | 6 | 8 | 4 | 9 | 4 | 4 | 4 | 4
Completed | 4 | 6 | 8 | 4 | 9 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A Group 1 Cohort 1: Single Dose IV Tedizolid Phosphate 28 Days to <6 Months | Part A Group 1 Cohort 2: Single Dose IV Tedizolid Phosphate 6 Months to <24 Months | Part A Group 2 Cohort 1: Single Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 2 Cohort 2: Multiple Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 3 Cohort 1: Single Dose IV Tedizolid Phosphate (Preterm) Birth to <28 Days | Part A Group 3 Cohort 2: Multiple Dose IV Tedizolid Phosphate IV (Preterm) Birth to <28 Days | Part B Group 4: Single Dose Oral Tedizolid Phosphate 28 Days to <24 Months | Part B Group 5: Single Dose Oral Tedizolid Phosphate (Full Term) Birth to <28 Days | Part B Group 6: Single Dose Oral Tedizolid Phosphate (Preterm) Birth to <28 Days | Total
Number analyzed (Participants) | 4 | 6 | 8 | 4 | 9 | 4 | 4 | 4 | 4 | 47
Age, Continuous [Mean (Standard Deviation); unit: Days] | 51.3 (9.9) | 420.7 (167.1) | 8.3 (9.4) | 11.8 (11.3) | 9.9 (7.9) | 2.0 (1.2) | 289.0 (165.5) | 13.0 (11.7) | 6.5 (6.4) | 88.8 (165.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 5 | 1 | 3 | 2 | 2 | 0 | 1 | 18
  Male | 2 | 4 | 3 | 3 | 6 | 2 | 2 | 4 | 3 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 7 | 3 | 3 | 2 | 0 | 2 | 3 | 20
  Not Hispanic or Latino | 4 | 6 | 1 | 1 | 5 | 2 | 4 | 2 | 1 | 26
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  White | 3 | 5 | 2 | 1 | 6 | 2 | 4 | 2 | 1 | 26
  More than one race | 0 | 1 | 6 | 2 | 3 | 2 | 0 | 2 | 3 | 19
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part A: Area Under the Concentration-time Curve From Time 0 to Time of Last Quantifiable Drug Concentration (AUC0-last) of Tedizolid Phosphate (Prodrug) After Single-dose IV Administration
Description: AUC0-last of tedizolid phosphate was quantified in participants receiving tedizolid phosphate. Protocol specified analysis of pharmacokinetic (PK) outcomes in Group 1 was done irrespective of age (28 days to <24 months, across ages in Cohorts 1 and 2). As specified in the protocol, tedizolid phosphate AUC0-last for multiple dose (Part A Group 2 Cohort 2, Group 3 Cohort 2) were not included in this outcome and have been reported separately in the record. Tedizolid phosphate PK analysis was not planned or conducted in Part B (Groups 4, 5, 6), per protocol.
Time Frame: 1, 1.5, 3, 6, 12 and 24 hours post start of dosing
Population: The subset of participants who complied with the protocol to ensure that data would exhibit treatment effects, according to the scientific model and had data available for this outcome. Per protocol, Group 1 PK outcome analysis was done irrespective of age, across Cohorts 1 and 2 (28 days to <24 months). AUC0-last for multiple dose (Part A Group 2 Cohort 2, Group 3 Cohort 2) are excluded and have been reported separately. Tedizolid phosphate PK analysis was not done in Part B, per protocol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*μg/mL
Groups:
- Group 1 Cohorts 1+2:SD IV Tedizolid Phosphate 28days-<24months: Pediatric participants 28 days to <24 months of age received a single dose (SD) intravenous (IV) infusion of tedizolid phosphate according to body weight: 3 mg/kg for body weight <10 kg or 2.5 mg/kg for body weight 10 to <30 kg.
Arm/Group | Group 1 Cohorts 1+2:SD IV Tedizolid Phosphate 28days-<24months | Part A Group 2 Cohort 1: Single Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 2 Cohort 2: Multiple Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 3 Cohort 1: Single Dose IV Tedizolid Phosphate (Preterm) Birth to <28 Days | Part A Group 3 Cohort 2: Multiple Dose IV Tedizolid Phosphate IV (Preterm) Birth to <28 Days | Part B Group 4: Single Dose Oral Tedizolid Phosphate 28 Days to <24 Months | Part B Group 5: Single Dose Oral Tedizolid Phosphate (Full Term) Birth to <28 Days | Part B Group 6: Single Dose Oral Tedizolid Phosphate (Preterm) Birth to <28 Days
Number analyzed (Participants) | 3 | 1 | 0 | 3 | 0 | 0 | 0 | 0
hr*μg/mL | NA (NA) — Measure type and method of dispersion could not be estimated per protocol due to plasma concentrations below level of quantification (BLOQ). | NA (NA) — Measure type could not be estimated per protocol due to plasma concentrations BLOQ. Method of dispersion not applicable due to low number of participants analyzed. |  | NA (NA) — Measure type and method of dispersion could not be estimated per protocol due to plasma concentrations below level of quantification (BLOQ). |  |  |  |

2. Primary Outcome: Part A: Area Under the Concentration-time Curve From Time 0 to Infinity (AUC0-inf) of Tedizolid Phosphate (Prodrug) After Single-dose IV Administration
Description: AUC0-inf of tedizolid phosphate was quantified in participants receiving tedizolid phosphate. Protocol specified analysis of PK outcomes in Group 1 was done irrespective of age (28 days to <24 months, across ages in Cohorts 1 and 2). As specified in the protocol, tedizolid phosphate AUC0-inf for multiple dose (Part A Group 2 Cohort 2, Group 3 Cohort 2) were not included in this outcome and have been reported separately in the record. Tedizolid phosphate PK analysis was not planned or conducted in Part B (Groups 4, 5, 6), per protocol.
Time Frame: 1, 1.5, 3, 6, 12 and 24 hours post start of dosing
Population: The subset of participants who complied with the protocol to ensure that data would exhibit treatment effects, according to the scientific model and had data available for this outcome. Per protocol, Group 1 PK outcome analysis was done irrespective of age, across Cohorts 1 and 2 (28 days to <24 months). AUC0-inf for multiple dose (Part A Group 2 Cohort 2, Group 3 Cohort 2) are excluded and have been reported separately. Tedizolid phosphate PK analysis was not done in Part B, per protocol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*μg/mL
Arm/Group | Group 1 Cohorts 1+2:SD IV Tedizolid Phosphate 28days-<24months | Part A Group 2 Cohort 1: Single Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 2 Cohort 2: Multiple Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 3 Cohort 1: Single Dose IV Tedizolid Phosphate (Preterm) Birth to <28 Days | Part A Group 3 Cohort 2: Multiple Dose IV Tedizolid Phosphate IV (Preterm) Birth to <28 Days | Part B Group 4: Single Dose Oral Tedizolid Phosphate 28 Days to <24 Months | Part B Group 5: Single Dose Oral Tedizolid Phosphate (Full Term) Birth to <28 Days | Part B Group 6: Single Dose Oral Tedizolid Phosphate (Preterm) Birth to <28 Days
Number analyzed (Participants) | 3 | 1 | 0 | 3 | 0 | 0 | 0 | 0
hr*μg/mL | NA (NA) — Measure type and method of dispersion could not be estimated per protocol due to plasma concentrations BLOQ. | NA (NA) — Measure type could not be estimated per protocol due to plasma concentrations BLOQ. Method of dispersion not applicable due to low number of participants analyzed. |  | NA (NA) — Measure type and method of dispersion could not be estimated per protocol due to plasma concentrations BLOQ. |  |  |  |

3. Primary Outcome: Part A: Maximum Concentration (Cmax) of Tedizolid Phosphate (Prodrug) After Single-dose IV Administration
Description: Cmax of tedizolid phosphate was quantified in participants receiving tedizolid phosphate. Protocol specified analysis of PK outcomes in Group 1 was done irrespective of age (28 days to <24 months, across ages in Cohorts 1 and 2). As specified in the protocol, tedizolid phosphate Cmax for multiple dose (Part A Group 2 Cohort 2, Group 3 Cohort 2) were not included in this outcome and have been reported separately in the record. Tedizolid phosphate PK analysis was not planned or conducted in Part B (Groups 4, 5, 6), per protocol.
Time Frame: 1, 1.5, 3, 6, 12 and 24 hours post start of dosing
Population: The subset of participants who complied with the protocol to ensure that data would exhibit treatment effects, according to the scientific model and had data available for this outcome. Per protocol, Group 1 PK outcome analysis was done irrespective of age, across Cohorts 1 and 2 (28 days to <24 months). Cmax for multiple dose (Part A Group 2 Cohort 2, Group 3 Cohort 2) are excluded and have been reported separately. Tedizolid phosphate PK analysis was not done in Part B, per protocol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Group 1 Cohorts 1+2:SD IV Tedizolid Phosphate 28days-<24months | Part A Group 2 Cohort 1: Single Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 2 Cohort 2: Multiple Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 3 Cohort 1: Single Dose IV Tedizolid Phosphate (Preterm) Birth to <28 Days | Part A Group 3 Cohort 2: Multiple Dose IV Tedizolid Phosphate IV (Preterm) Birth to <28 Days | Part B Group 4: Single Dose Oral Tedizolid Phosphate 28 Days to <24 Months | Part B Group 5: Single Dose Oral Tedizolid Phosphate (Full Term) Birth to <28 Days | Part B Group 6: Single Dose Oral Tedizolid Phosphate (Preterm) Birth to <28 Days
Number analyzed (Participants) | 3 | 1 | 0 | 3 | 0 | 0 | 0 | 0
μg/mL | NA (NA) — Measure type and method of dispersion could not be estimated per protocol due to plasma concentrations BLOQ. | NA (NA) — Measure type could not be estimated per protocol due to plasma concentrations BLOQ. Method of dispersion not applicable due to low number of participants analyzed. |  | NA (NA) — Measure type and method of dispersion could not be estimated per protocol due to plasma concentrations BLOQ. |  |  |  |

4. Primary Outcome: Part A: Time to Reach Maximum Concentration (Tmax) of Tedizolid Phosphate (Prodrug) After Single-dose IV Administration
Description: Tmax of tedizolid phosphate was quantified in participants receiving tedizolid phosphate. Protocol specified analysis of PK outcomes in Group 1 was done irrespective of age (28 days to <24 months, across ages in Cohorts 1 and 2). As specified in the protocol, tedizolid phosphate Tmax for multiple dose (Part A Group 2 Cohort 2, Group 3 Cohort 2) were not included in this outcome and have been reported separately in the record. Tedizolid phosphate PK analysis was not planned or conducted in Part B (Groups 4, 5, 6), per protocol.
Time Frame: 1, 1.5, 3, 6, 12 and 24 hours post start of dosing
Population: The subset of participants who complied with the protocol to ensure that data would exhibit treatment effects, according to the scientific model and had data available for this outcome. Per protocol, Group 1 PK outcome analysis was done irrespective of age, across Cohorts 1 and 2 (28 days to <24 months). Tmax for multiple dose (Part A Group 2 Cohort 2, Group 3 Cohort 2) are excluded and have been reported separately. Tedizolid phosphate PK analysis was not done in Part B, per protocol.
Measure: Median (Full Range); unit: hr
Arm/Group | Group 1 Cohorts 1+2:SD IV Tedizolid Phosphate 28days-<24months | Part A Group 2 Cohort 1: Single Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 2 Cohort 2: Multiple Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 3 Cohort 1: Single Dose IV Tedizolid Phosphate (Preterm) Birth to <28 Days | Part A Group 3 Cohort 2: Multiple Dose IV Tedizolid Phosphate IV (Preterm) Birth to <28 Days | Part B Group 4: Single Dose Oral Tedizolid Phosphate 28 Days to <24 Months | Part B Group 5: Single Dose Oral Tedizolid Phosphate (Full Term) Birth to <28 Days | Part B Group 6: Single Dose Oral Tedizolid Phosphate (Preterm) Birth to <28 Days
Number analyzed (Participants) | 3 | 1 | 0 | 3 | 0 | 0 | 0 | 0
hr | NA [NA to NA] — Measure type and method of dispersion could not be estimated per protocol due to plasma concentrations BLOQ. | NA [NA to NA] — Measure type could not be estimated per protocol due to plasma concentrations BLOQ. Method of dispersion not applicable due to low number of participants analyzed. |  | NA [NA to NA] — Measure type and method of dispersion could not be estimated per protocol due to plasma concentrations BLOQ. |  |  |  |

5. Primary Outcome: Part A: Apparent Terminal Half-life (t½) of Tedizolid Phosphate (Prodrug) After Single-dose IV Administration
Description: t½ of tedizolid phosphate was quantified in participants receiving tedizolid phosphate. Protocol specified analysis of PK outcomes in Group 1 was done irrespective of age (28 days to <24 months, across ages in Cohorts 1 and 2). As specified in the protocol, tedizolid phosphate t½ for multiple dose (Part A Group 2 Cohort 2, Group 3 Cohort 2) were not included in this outcome and have been reported separately in the record. Tedizolid phosphate PK analysis was not planned or conducted in Part B (Groups 4, 5, 6), per protocol.
Time Frame: 1, 1.5, 3, 6, 12 and 24 hours post start of dosing
Population: The subset of participants who complied with the protocol to ensure that data would exhibit treatment effects, according to the scientific model and had data available for this outcome. Per protocol, Group 1 PK outcome analysis was done irrespective of age, across Cohorts 1 and 2 (28 days to <24 months). t1/2 for multiple dose (Part A Group 2 Cohort 2, Group 3 Cohort 2) are excluded and have been reported separately. Tedizolid phosphate PK analysis was not done in Part B, per protocol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Group 1 Cohorts 1+2:SD IV Tedizolid Phosphate 28days-<24months | Part A Group 2 Cohort 1: Single Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 2 Cohort 2: Multiple Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 3 Cohort 1: Single Dose IV Tedizolid Phosphate (Preterm) Birth to <28 Days | Part A Group 3 Cohort 2: Multiple Dose IV Tedizolid Phosphate IV (Preterm) Birth to <28 Days | Part B Group 4: Single Dose Oral Tedizolid Phosphate 28 Days to <24 Months | Part B Group 5: Single Dose Oral Tedizolid Phosphate (Full Term) Birth to <28 Days | Part B Group 6: Single Dose Oral Tedizolid Phosphate (Preterm) Birth to <28 Days
Number analyzed (Participants) | 3 | 1 | 0 | 3 | 0 | 0 | 0 | 0
hr | NA (NA) — Measure type and method of dispersion could not be estimated per protocol due to plasma concentrations BLOQ. | NA (NA) — Measure type could not be estimated per protocol due to plasma concentrations BLOQ. Method of dispersion not applicable due to low number of participants analyzed. |  | NA (NA) — Measure type and method of dispersion could not be estimated per protocol due to plasma concentrations BLOQ. |  |  |  |

6. Primary Outcome: Part A: AUC0-last of Tedizolid Phosphate (Prodrug) After Multiple-dose IV Administration
Description: AUC0-last of tedizolid phosphate was quantified in participants receiving tedizolid phosphate. As specified in the protocol, tedizolid phosphate AUC0-last for single dose (Part A Group 1 [Cohorts 1 and 2], Group 2 Cohort 1, Group 3 Cohort 1) were not included in this outcome and have been reported separately in the record. Tedizolid phosphate PK analysis was not planned or conducted in Part B (Groups 4, 5, 6), per protocol. Participants in Group 2 Cohort 2 study arm did not meet the criteria for PK per protocol analysis population for this outcome and were excluded from this protocol-specified analysis.
Time Frame: Day 3: pre-dose, 1, 1.5, 3, 6 and 12 hours post start of dosing
Population: The subset of participants who complied with the protocol to ensure that data exhibits treatment effects and had data available for this outcome. AUC0-last for single dose (Part A Group 1 [Cohorts 1 & 2], Group 2 Cohort 1, Group 3 Cohort 1) are excluded and have been reported separately. Tedizolid phosphate PK analysis was not done in Part B, per protocol. Group 2 Cohort 2 participants didn't meet the per protocol analysis population criteria and were excluded from this analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*μg/mL
Arm/Group | Group 1 Cohorts 1+2:SD IV Tedizolid Phosphate 28days-<24months | Part A Group 2 Cohort 1: Single Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 2 Cohort 2: Multiple Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 3 Cohort 1: Single Dose IV Tedizolid Phosphate (Preterm) Birth to <28 Days | Part A Group 3 Cohort 2: Multiple Dose IV Tedizolid Phosphate IV (Preterm) Birth to <28 Days | Part B Group 4: Single Dose Oral Tedizolid Phosphate 28 Days to <24 Months | Part B Group 5: Single Dose Oral Tedizolid Phosphate (Full Term) Birth to <28 Days | Part B Group 6: Single Dose Oral Tedizolid Phosphate (Preterm) Birth to <28 Days
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
hr*μg/mL |  |  |  |  | NA (NA) — Measure type and method of dispersion could not be estimated per protocol due to plasma concentrations BLOQ. |  |  |

7. Primary Outcome: Part A: AUC0-inf of Tedizolid Phosphate (Prodrug) After Multiple-dose IV Administration
Description: AUC0-inf of tedizolid phosphate was quantified in participants receiving tedizolid phosphate. As specified in the protocol, tedizolid phosphate AUC0-inf for single dose (Part A Group 1 [Cohorts 1 and 2], Group 2 Cohort 1, Group 3 Cohort 1) were not included in this outcome and have been reported separately in the record. Tedizolid phosphate PK analysis was not planned or conducted in Part B (Groups 4, 5, 6), per protocol. Participants in Group 2 Cohort 2 study arm did not meet the criteria for PK per protocol analysis population for this endpoint and were excluded from this protocol-specified analysis.
Time Frame: Day 3: pre-dose, 1, 1.5, 3, 6 and 12 hours post start of dosing
Population: The subset of participants who complied with the protocol to ensure that data exhibits treatment effects and had data available for this outcome. AUC0-inf for single dose (Part A Group 1 [Cohorts 1 & 2], Group 2 Cohort 1, Group 3 Cohort 1) are excluded and have been reported separately. Tedizolid phosphate PK analysis was not done in Part B, per protocol. Group 2 Cohort 2 participants didn't meet the per protocol analysis population criteria and were excluded from this analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*μg/mL
Arm/Group | Group 1 Cohorts 1+2:SD IV Tedizolid Phosphate 28days-<24months | Part A Group 2 Cohort 1: Single Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 2 Cohort 2: Multiple Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 3 Cohort 1: Single Dose IV Tedizolid Phosphate (Preterm) Birth to <28 Days | Part A Group 3 Cohort 2: Multiple Dose IV Tedizolid Phosphate IV (Preterm) Birth to <28 Days | Part B Group 4: Single Dose Oral Tedizolid Phosphate 28 Days to <24 Months | Part B Group 5: Single Dose Oral Tedizolid Phosphate (Full Term) Birth to <28 Days | Part B Group 6: Single Dose Oral Tedizolid Phosphate (Preterm) Birth to <28 Days
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
hr*μg/mL |  |  |  |  | NA (NA) — Measure type and method of dispersion could not be estimated per protocol due to plasma concentrations BLOQ. |  |  |

8. Primary Outcome: Part A: Cmax of Tedizolid Phosphate (Prodrug) After Multiple-dose IV Administration
Description: Cmax of tedizolid phosphate was quantified in participants receiving tedizolid phosphate. As specified in the protocol, tedizolid phosphate Cmax for single dose (Part A Group 1 [Cohorts 1 and 2], Group 2 Cohort 1, Group 3 Cohort 1) were not included in this outcome and have been reported separately in the record. Tedizolid phosphate PK analysis was not planned or conducted in Part B (Groups 4, 5, 6), per protocol. Participants in Group 2 Cohort 2 study arm did not meet the criteria for PK per protocol analysis population for this outcome and were excluded from this protocol-specified analysis.
Time Frame: Day 3: pre-dose, 1, 1.5, 3, 6 and 12 hours post start of dosing
Population: The subset of participants who complied with the protocol to ensure that data exhibits treatment effects and had data available for this outcome. Cmax for single dose (Part A Group 1 [Cohorts 1 & 2], Group 2 Cohort 1, Group 3 Cohort 1) are excluded and have been reported separately. Tedizolid phosphate PK analysis was not done in Part B, per protocol. Group 2 Cohort 2 participants didn't meet the per protocol analysis population criteria and were excluded from this analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Group 1 Cohorts 1+2:SD IV Tedizolid Phosphate 28days-<24months | Part A Group 2 Cohort 1: Single Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 2 Cohort 2: Multiple Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 3 Cohort 1: Single Dose IV Tedizolid Phosphate (Preterm) Birth to <28 Days | Part A Group 3 Cohort 2: Multiple Dose IV Tedizolid Phosphate IV (Preterm) Birth to <28 Days | Part B Group 4: Single Dose Oral Tedizolid Phosphate 28 Days to <24 Months | Part B Group 5: Single Dose Oral Tedizolid Phosphate (Full Term) Birth to <28 Days | Part B Group 6: Single Dose Oral Tedizolid Phosphate (Preterm) Birth to <28 Days
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
μg/mL |  |  |  |  | NA (NA) — Measure type and method of dispersion could not be estimated per protocol due to plasma concentrations BLOQ. |  |  |

9. Primary Outcome: Part A: Tmax of Tedizolid Phosphate (Prodrug) After Multiple-dose IV Administration
Description: Tmax of tedizolid phosphate was quantified in participants receiving tedizolid phosphate. As specified in the protocol, tedizolid phosphate Tmax for single dose (Part A Group 1 [Cohorts 1 and 2], Group 2 Cohort 1, Group 3 Cohort 1) were not included in this outcome and have been reported separately in the record. Tedizolid phosphate PK analysis was not planned or conducted in Part B (Groups 4, 5, 6), per protocol. Participants in Group 2 Cohort 2 study arm did not meet the criteria for PK per protocol analysis population for this outcome and were excluded from this protocol-specified analysis.
Time Frame: Day 3: pre-dose, 1, 1.5, 3, 6 and 12 hours post start of dosing
Population: The subset of participants who complied with the protocol to ensure that data exhibits treatment effects and had data available for this outcome. Tmax for single dose (Part A Group 1 [Cohorts 1 & 2], Group 2 Cohort 1, Group 3 Cohort 1) are excluded and have been reported separately. Tedizolid phosphate PK analysis was not done in Part B, per protocol. Group 2 Cohort 2 participants didn't meet the per protocol analysis population criteria and were excluded from this analysis.
Measure: Median (Full Range); unit: hr
Arm/Group | Group 1 Cohorts 1+2:SD IV Tedizolid Phosphate 28days-<24months | Part A Group 2 Cohort 1: Single Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 2 Cohort 2: Multiple Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 3 Cohort 1: Single Dose IV Tedizolid Phosphate (Preterm) Birth to <28 Days | Part A Group 3 Cohort 2: Multiple Dose IV Tedizolid Phosphate IV (Preterm) Birth to <28 Days | Part B Group 4: Single Dose Oral Tedizolid Phosphate 28 Days to <24 Months | Part B Group 5: Single Dose Oral Tedizolid Phosphate (Full Term) Birth to <28 Days | Part B Group 6: Single Dose Oral Tedizolid Phosphate (Preterm) Birth to <28 Days
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
hr |  |  |  |  | NA [NA to NA] — Measure type and method of dispersion could not be estimated per protocol due to plasma concentrations BLOQ. |  |  |

10. Primary Outcome: Part A: t½ of Tedizolid Phosphate (Prodrug) After Multiple-dose IV Administration
Description: t½ of tedizolid phosphate was quantified in participants receiving tedizolid phosphate. As specified in the protocol, tedizolid phosphate t½ for single dose (Part A Group 1 [Cohorts 1 and 2], Group 2 Cohort 1, Group 3 Cohort 1) were not included in this outcome and have been reported separately in the record. Tedizolid phosphate PK analysis was not planned or conducted in Part B (Groups 4, 5, 6), per protocol. Participants in Group 2 Cohort 2 study arm did not meet the criteria for PK per protocol analysis population for this outcome and were excluded from this protocol-specified analysis.
Time Frame: Day 3: pre-dose, 1, 1.5, 3, 6 and 12 hours post start of dosing
Population: The subset of participants who complied with the protocol to ensure that data exhibits treatment effects and had data available for this outcome. t1/2 for single dose (Part A Group 1 [Cohorts 1 & 2], Group 2 Cohort 1, Group 3 Cohort 1) are excluded and have been reported separately. Tedizolid phosphate PK analysis was not done in Part B, per protocol. Group 2 Cohort 2 participants didn't meet the per protocol analysis population criteria and were excluded from this analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Group 1 Cohorts 1+2:SD IV Tedizolid Phosphate 28days-<24months | Part A Group 2 Cohort 1: Single Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 2 Cohort 2: Multiple Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 3 Cohort 1: Single Dose IV Tedizolid Phosphate (Preterm) Birth to <28 Days | Part A Group 3 Cohort 2: Multiple Dose IV Tedizolid Phosphate IV (Preterm) Birth to <28 Days | Part B Group 4: Single Dose Oral Tedizolid Phosphate 28 Days to <24 Months | Part B Group 5: Single Dose Oral Tedizolid Phosphate (Full Term) Birth to <28 Days | Part B Group 6: Single Dose Oral Tedizolid Phosphate (Preterm) Birth to <28 Days
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
hr |  |  |  |  | NA (NA) — Measure type and method of dispersion could not be estimated per protocol due to plasma concentrations BLOQ. |  |  |

11. Primary Outcome: Part A: AUC0-24 of Tedizolid (Active Metabolite) After Single-dose IV Administration of Tedizolid Phosphate [AUC0-last]
Description: AUC0-last of tedizolid (metabolite) was quantified in participants receiving tedizolid phosphate. Protocol specified analysis of PK endpoints in Group 1 was done irrespective of age (28 days to <24 months, across ages in Cohorts 1 and 2). As specified in the protocol, AUC0-last for tedizolid metabolite in multiple dose (Part A Group 2 Cohort 2, Group 3 Cohort 2) and Part B (Groups 4, 5, 6) were not included in this endpoint and have been reported separately in the record.
Time Frame: 1, 1.5, 3, 6, 12 and 24 hours post start of dosing
Population: The subset of participants who complied with the protocol to ensure that data would exhibit treatment effects, according to the scientific model and had data available for this outcome. Per protocol, Group 1 PK outcome analysis was done irrespective of age, across Cohorts 1 and 2 (28 days to <24 months). AUC0-last for multiple dose (Part A Group 2 Cohort 2, Group 3 Cohort 2) and Part B (Groups 4, 5, 6) are excluded and have been reported separately.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*μg/mL
Arm/Group | Group 1 Cohorts 1+2:SD IV Tedizolid Phosphate 28days-<24months | Part A Group 2 Cohort 1: Single Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 2 Cohort 2: Multiple Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 3 Cohort 1: Single Dose IV Tedizolid Phosphate (Preterm) Birth to <28 Days | Part A Group 3 Cohort 2: Multiple Dose IV Tedizolid Phosphate IV (Preterm) Birth to <28 Days | Part B Group 4: Single Dose Oral Tedizolid Phosphate 28 Days to <24 Months | Part B Group 5: Single Dose Oral Tedizolid Phosphate (Full Term) Birth to <28 Days | Part B Group 6: Single Dose Oral Tedizolid Phosphate (Preterm) Birth to <28 Days
Number analyzed (Participants) | 10 | 5 | 0 | 3 | 0 | 0 | 0 | 0
hr*μg/mL | 13.6 (42.4) | 8.23 (115.9) |  | 15.6 (17.6) |  |  |  |

12. Primary Outcome: Part A: AUC0-inf of Tedizolid (Active Metabolite) After Single-dose IV Administration of Tedizolid Phosphate
Description: AUC0-inf of tedizolid (metabolite) was quantified in participants receiving tedizolid phosphate. Protocol specified analysis of PK endpoints in Group 1 was done irrespective of age (28 days to <24 months, across ages in Cohorts 1 and 2). As specified in the protocol, AUC0-inf for tedizolid metabolite in multiple dose (Part A Group 2 Cohort 2, Group 3 Cohort 2) and Part B (Groups 4, 5, 6) were not included in this endpoint and have been reported separately in the record.
Time Frame: 1, 1.5, 3, 6, 12 and 24 hours post start of dosing
Population: The subset of participants who complied with the protocol to ensure that data would exhibit treatment effects, according to the scientific model and had data available for this outcome. Per protocol, Group 1 PK outcome analysis was done irrespective of age, across Cohorts 1 and 2 (28 days to <24 months). AUC0-inf for multiple dose (Part A Group 2 Cohort 2, Group 3 Cohort 2) and Part B (Groups 4, 5, 6) are excluded and have been reported separately.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*μg/mL
Arm/Group | Group 1 Cohorts 1+2:SD IV Tedizolid Phosphate 28days-<24months | Part A Group 2 Cohort 1: Single Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 2 Cohort 2: Multiple Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 3 Cohort 1: Single Dose IV Tedizolid Phosphate (Preterm) Birth to <28 Days | Part A Group 3 Cohort 2: Multiple Dose IV Tedizolid Phosphate IV (Preterm) Birth to <28 Days | Part B Group 4: Single Dose Oral Tedizolid Phosphate 28 Days to <24 Months | Part B Group 5: Single Dose Oral Tedizolid Phosphate (Full Term) Birth to <28 Days | Part B Group 6: Single Dose Oral Tedizolid Phosphate (Preterm) Birth to <28 Days
Number analyzed (Participants) | 10 | 5 | 0 | 3 | 0 | 0 | 0 | 0
hr*μg/mL | 14.3 (40.4) | 9.21 (128.2) |  | 17.8 (20.9) |  |  |  |

13. Primary Outcome: Part A: Cmax of Tedizolid (Active Metabolite) After Single-dose IV Administration of Tedizolid Phosphate
Description: Cmax of tedizolid (metabolite) was quantified in participants receiving tedizolid phosphate. Protocol specified analysis of PK endpoints in Group 1 was done irrespective of age (28 days to <24 months, across ages in Cohorts 1 and 2). As specified in the protocol, Cmax for tedizolid metabolite in multiple dose (Part A Group 2 Cohort 2, Group 3 Cohort 2) and Part B (Groups 4, 5, 6) were not included in this endpoint and have been reported separately in the record.
Time Frame: 1, 1.5, 3, 6, 12 and 24 hours post start of dosing
Population: The subset of participants who complied with the protocol to ensure that data would exhibit treatment effects, according to the scientific model and had data available for this outcome. Per protocol, Group 1 PK outcome analysis was done irrespective of age, across Cohorts 1 and 2 (28 days to <24 months). Cmax for multiple dose (Part A Group 2 Cohort 2, Group 3 Cohort 2) and Part B (Groups 4, 5, 6) are excluded and have been reported separately.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Group 1 Cohorts 1+2:SD IV Tedizolid Phosphate 28days-<24months | Part A Group 2 Cohort 1: Single Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 2 Cohort 2: Multiple Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 3 Cohort 1: Single Dose IV Tedizolid Phosphate (Preterm) Birth to <28 Days | Part A Group 3 Cohort 2: Multiple Dose IV Tedizolid Phosphate IV (Preterm) Birth to <28 Days | Part B Group 4: Single Dose Oral Tedizolid Phosphate 28 Days to <24 Months | Part B Group 5: Single Dose Oral Tedizolid Phosphate (Full Term) Birth to <28 Days | Part B Group 6: Single Dose Oral Tedizolid Phosphate (Preterm) Birth to <28 Days
Number analyzed (Participants) | 10 | 6 | 0 | 5 | 0 | 0 | 0 | 0
μg/mL | 2.19 (51.0) | 0.962 (71.9) |  | 1.35 (44.5) |  |  |  |

14. Primary Outcome: Part A: Tmax of Tedizolid (Active Metabolite) After Single-dose IV Administration of Tedizolid Phosphate
Description: Tmax of tedizolid (metabolite) was quantified in participants receiving tedizolid phosphate. Protocol specified analysis of PK endpoints in Group 1 was done irrespective of age (28 days to <24 months, across ages in Cohorts 1 and 2). As specified in the protocol, Tmax for tedizolid metabolite in multiple dose (Part A Group 2 Cohort 2, Group 3 Cohort 2) and Part B (Groups 4, 5, 6) were not included in this endpoint and have been reported separately in the record.
Time Frame: 1, 1.5, 3, 6, 12 and 24 hours post start of dosing
Population: The subset of participants who complied with the protocol to ensure that data would exhibit treatment effects, according to the scientific model and had data available for this outcome. Per protocol, Group 1 PK outcome analysis was done irrespective of age, across Cohorts 1 and 2 (28 days to <24 months). Tmax for multiple dose (Part A Group 2 Cohort 2, Group 3 Cohort 2) and Part B (Groups 4, 5, 6) are excluded and have been reported separately.
Measure: Median (Full Range); unit: hr
Arm/Group | Group 1 Cohorts 1+2:SD IV Tedizolid Phosphate 28days-<24months | Part A Group 2 Cohort 1: Single Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 2 Cohort 2: Multiple Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 3 Cohort 1: Single Dose IV Tedizolid Phosphate (Preterm) Birth to <28 Days | Part A Group 3 Cohort 2: Multiple Dose IV Tedizolid Phosphate IV (Preterm) Birth to <28 Days | Part B Group 4: Single Dose Oral Tedizolid Phosphate 28 Days to <24 Months | Part B Group 5: Single Dose Oral Tedizolid Phosphate (Full Term) Birth to <28 Days | Part B Group 6: Single Dose Oral Tedizolid Phosphate (Preterm) Birth to <28 Days
Number analyzed (Participants) | 10 | 6 | 0 | 5 | 0 | 0 | 0 | 0
hr | 1.33 [1.00 to 1.58] | 1.41 [1.00 to 2.50] |  | 1.50 [1.08 to 6.53] |  |  |  |

15. Primary Outcome: Part A: t½ of Tedizolid (Active Metabolite) After Single-dose IV Administration of Tedizolid Phosphate
Description: t½ of tedizolid (metabolite) was quantified in participants receiving tedizolid phosphate. Protocol specified analysis of PK endpoints in Group 1 was done irrespective of age (28 days to <24 months, across ages in Cohorts 1 and 2). As specified in the protocol, t½ for tedizolid metabolite in multiple dose (Part A Group 2 Cohort 2, Group 3 Cohort 2) and Part B (Groups 4, 5, 6) were not included in this endpoint and have been reported separately in the record.
Time Frame: 1, 1.5, 3, 6, 12 and 24 hours post start of dosing
Population: The subset of participants who complied with the protocol to ensure that data would exhibit treatment effects, according to the scientific model and had data available for this outcome. Per protocol, Group 1 PK outcome analysis was done irrespective of age, across Cohorts 1 and 2 (28 days to <24 months). t1/2 for multiple dose (Part A Group 2 Cohort 2, Group 3 Cohort 2) and Part B (Groups 4, 5, 6) are excluded and have been reported separately.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Group 1 Cohorts 1+2:SD IV Tedizolid Phosphate 28days-<24months | Part A Group 2 Cohort 1: Single Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 2 Cohort 2: Multiple Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 3 Cohort 1: Single Dose IV Tedizolid Phosphate (Preterm) Birth to <28 Days | Part A Group 3 Cohort 2: Multiple Dose IV Tedizolid Phosphate IV (Preterm) Birth to <28 Days | Part B Group 4: Single Dose Oral Tedizolid Phosphate 28 Days to <24 Months | Part B Group 5: Single Dose Oral Tedizolid Phosphate (Full Term) Birth to <28 Days | Part B Group 6: Single Dose Oral Tedizolid Phosphate (Preterm) Birth to <28 Days
Number analyzed (Participants) | 10 | 5 | 0 | 3 | 0 | 0 | 0 | 0
hr | 4.17 (47.7) | 6.63 (38.0) |  | 7.08 (41.2) |  |  |  |

16. Primary Outcome: Part A: AUC0-12 of Tedizolid (Active Metabolite) After Multiple-dose IV Administration of Tedizolid Phosphate [AUC0-last]
Description: AUC0-last of tedizolid (metabolite) was quantified in participants receiving tedizolid phosphate. The per protocol statistical approach used in this noncompartmental analysis allowed data collected to generate single concentration listing. This was analyzed in the per protocol population consisting of the subset of participants who complied with the protocol sufficiently to ensure that these data would be likely to exhibit treatment effects, based on the underlying scientific model and had data available for this endpoint. As specified in the protocol, AUC0-last for tedizolid metabolite in single dose (Part A Group 1 [Cohorts 1 and 2], Group 2 Cohort 1, Group 3 Cohort 1; Part B [Groups 4, 5, 6]) were not included in this endpoint and have been reported separately in the record.
Time Frame: Day 3: pre-dose, 1, 1.5, 3, 6 and 12 hours post start of dosing
Population: The subset of participants who complied with protocol to ensure that data exhibits treatment effects, according to scientific model and had data available for this outcome. AUC0-last for tedizolid metabolite in single dose (Part A Group 1 [Cohorts 1 and 2], Group 2 Cohort 1, Group 3 Cohort 1; Part B [Groups 4, 5, 6]) are excluded and have been reported separately.
Measure: Number; unit: hr*μg/mL
Arm/Group | Group 1 Cohorts 1+2:SD IV Tedizolid Phosphate 28days-<24months | Part A Group 2 Cohort 1: Single Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 2 Cohort 2: Multiple Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 3 Cohort 1: Single Dose IV Tedizolid Phosphate (Preterm) Birth to <28 Days | Part A Group 3 Cohort 2: Multiple Dose IV Tedizolid Phosphate IV (Preterm) Birth to <28 Days | Part B Group 4: Single Dose Oral Tedizolid Phosphate 28 Days to <24 Months | Part B Group 5: Single Dose Oral Tedizolid Phosphate (Full Term) Birth to <28 Days | Part B Group 6: Single Dose Oral Tedizolid Phosphate (Preterm) Birth to <28 Days
Number analyzed (Participants) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
hr*μg/mL |  |  | 10.5 |  | 7.48 |  |  |

17. Primary Outcome: Part A: Cmax of Tedizolid (Active Metabolite) After Multiple-dose IV Administration of Tedizolid Phosphate
Description: Cmax of tedizolid (metabolite) was quantified in participants receiving tedizolid phosphate. The per protocol statistical approach used in this noncompartmental analysis allowed data collected to generate single concentration listing. As specified in the protocol, Cmax for tedizolid metabolite in single dose (Part A Group 1 [Cohorts 1 and 2], Group 2 Cohort 1, Group 3 Cohort 1; Part B [Groups 4, 5, 6]) were not included in this endpoint and have been reported separately in the record.
Time Frame: Day 3: pre-dose, 1, 1.5, 3, 6 and 12 hours post start of dosing
Population: The subset of participants who complied with protocol to ensure that data exhibits treatment effects, according to scientific model and had data available for this outcome. Cmax for tedizolid metabolite in single dose (Part A Group 1 [Cohorts 1 and 2], Group 2 Cohort 1, Group 3 Cohort 1; Part B [Groups 4, 5, 6]) are excluded and have been reported separately.
Measure: Number; unit: μg/mL
Arm/Group | Group 1 Cohorts 1+2:SD IV Tedizolid Phosphate 28days-<24months | Part A Group 2 Cohort 1: Single Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 2 Cohort 2: Multiple Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 3 Cohort 1: Single Dose IV Tedizolid Phosphate (Preterm) Birth to <28 Days | Part A Group 3 Cohort 2: Multiple Dose IV Tedizolid Phosphate IV (Preterm) Birth to <28 Days | Part B Group 4: Single Dose Oral Tedizolid Phosphate 28 Days to <24 Months | Part B Group 5: Single Dose Oral Tedizolid Phosphate (Full Term) Birth to <28 Days | Part B Group 6: Single Dose Oral Tedizolid Phosphate (Preterm) Birth to <28 Days
Number analyzed (Participants) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
μg/mL |  |  | 1.82 |  | 1.69 |  |  |

18. Primary Outcome: Part A: Tmax of Tedizolid (Active Metabolite) After Multiple-dose IV Administration of Tedizolid Phosphate
Description: Tmax of tedizolid (metabolite) was quantified in participants receiving tedizolid phosphate. The per protocol statistical approach used in this noncompartmental analysis allowed data collected to generate single listing. As specified in the protocol, Tmax for tedizolid metabolite in single dose (Part A Group 1 [Cohorts 1 and 2], Group 2 Cohort 1, Group 3 Cohort 1; Part B [Groups 4, 5, 6]) were not included in this endpoint and have been reported separately in the record.
Time Frame: Day 3: pre-dose, 1, 1.5, 3, 6 and 12 hours post start of dosing
Population: The subset of participants who complied with protocol to ensure that data exhibits treatment effects, according to scientific model and had data available for this outcome. Tmax for tedizolid metabolite in single dose (Part A Group 1 [Cohorts 1 and 2], Group 2 Cohort 1, Group 3 Cohort 1; Part B [Groups 4, 5, 6]) are excluded and have been reported separately.
Measure: Number; unit: hr
Arm/Group | Group 1 Cohorts 1+2:SD IV Tedizolid Phosphate 28days-<24months | Part A Group 2 Cohort 1: Single Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 2 Cohort 2: Multiple Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 3 Cohort 1: Single Dose IV Tedizolid Phosphate (Preterm) Birth to <28 Days | Part A Group 3 Cohort 2: Multiple Dose IV Tedizolid Phosphate IV (Preterm) Birth to <28 Days | Part B Group 4: Single Dose Oral Tedizolid Phosphate 28 Days to <24 Months | Part B Group 5: Single Dose Oral Tedizolid Phosphate (Full Term) Birth to <28 Days | Part B Group 6: Single Dose Oral Tedizolid Phosphate (Preterm) Birth to <28 Days
Number analyzed (Participants) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
hr |  |  | 1.60 |  | 1.08 |  |  |

19. Primary Outcome: Part A: AUC0-inf of Tedizolid (Active Metabolite) After Multiple-dose IV Administration of Tedizolid Phosphate
Description: AUC0-inf of tedizolid (metabolite) was quantified in participants receiving tedizolid phosphate. The per protocol statistical approach to be used in this noncompartmental analysis would allow data collected to generate single concentration listing. However, protocol-specified PK sampling did not characterize the terminal elimination phase; therefore, AUC0-inf of tedizolid metabolite could not be estimated for multiple dose study arms (Part A Group 2 Cohort 2 and Part A Group 3 Cohort 2). As specified in the protocol, AUC0-inf for tedizolid metabolite in single dose (Part A Group 1[Cohorts 1 and 2],Group 2 Cohort 1, Group 3 Cohort 1; Part B[Groups 4, 5, 6]) were not included in this endpoint and have been reported separately in the record.
Time Frame: Day 3: pre-dose, 1, 1.5, 3, 6 and 12 hours post start of dosing
Population: The subset of participants who complied with protocol to ensure that data exhibits treatment effects, according to the scientific model. Protocol specified PK sampling didn't characterize terminal elimination phase; thus, this couldn't be estimated for multiple dose (Part A Group 2 Cohort 2, Group 3 Cohort 2). AUC0-inf for tedizolid metabolite in single dose (Part A Group 1 [Cohorts 1 and 2], Group 2 Cohort 1, Group 3 Cohort 1; Part B [Groups 4, 5, 6]) are excluded and reported separately.
Arm/Group | Group 1 Cohorts 1+2:SD IV Tedizolid Phosphate 28days-<24months | Part A Group 2 Cohort 1: Single Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 2 Cohort 2: Multiple Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 3 Cohort 1: Single Dose IV Tedizolid Phosphate (Preterm) Birth to <28 Days | Part A Group 3 Cohort 2: Multiple Dose IV Tedizolid Phosphate IV (Preterm) Birth to <28 Days | Part B Group 4: Single Dose Oral Tedizolid Phosphate 28 Days to <24 Months | Part B Group 5: Single Dose Oral Tedizolid Phosphate (Full Term) Birth to <28 Days | Part B Group 6: Single Dose Oral Tedizolid Phosphate (Preterm) Birth to <28 Days
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

20. Primary Outcome: Part A: t½ of Tedizolid (Active Metabolite) After Multiple-dose IV Administration of Tedizolid Phosphate
Description: t½ of tedizolid (metabolite) was quantified in participants receiving tedizolid phosphate. The per protocol statistical approach to be used in this noncompartmental analysis would allow data collected to generate single listing. However, protocol-specified PK sampling did not characterize the terminal elimination phase; therefore, t½ could not be estimated for multiple dose study arms (Part A Group 2 Cohort 2 and Part A Group 3 Cohort 2). As specified in the protocol, t½ for tedizolid metabolite in single dose (Part A Group 1 [Cohorts 1 and 2], Group 2 Cohort 1, Group 3 Cohort 1; Part B [Groups 4, 5, 6]) were not included in this endpoint and have been reported separately in the record.
Time Frame: Day 3: pre-dose, 1, 1.5, 3, 6 and 12 hours post start of dosing
Population: The subset of participants who complied with protocol to ensure that data exhibits treatment effects, according to the scientific model. Protocol specified PK sampling didn't characterize terminal elimination phase; thus, this couldn't be estimated for multiple dose (Part A Group 2 Cohort 2, Group 3 Cohort 2). t1/2 for tedizolid metabolite in single dose (Part A Group 1 [Cohorts 1 and 2], Group 2 Cohort 1, Group 3 Cohort 1; Part B [Groups 4, 5, 6]) are excluded and reported separately.
Arm/Group | Group 1 Cohorts 1+2:SD IV Tedizolid Phosphate 28days-<24months | Part A Group 2 Cohort 1: Single Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 2 Cohort 2: Multiple Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 3 Cohort 1: Single Dose IV Tedizolid Phosphate (Preterm) Birth to <28 Days | Part A Group 3 Cohort 2: Multiple Dose IV Tedizolid Phosphate IV (Preterm) Birth to <28 Days | Part B Group 4: Single Dose Oral Tedizolid Phosphate 28 Days to <24 Months | Part B Group 5: Single Dose Oral Tedizolid Phosphate (Full Term) Birth to <28 Days | Part B Group 6: Single Dose Oral Tedizolid Phosphate (Preterm) Birth to <28 Days
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

21. Primary Outcome: Part B: Area Under the Concentration-time Curve From Time 0 to 24 Hours (AUC0-24) of Tedizolid (Active Metabolite) After Single-dose Administration of Tedizolid Phosphate Oral Suspension [AUC0-last]
Description: AUC0-last of tedizolid (metabolite) was quantified in participants receiving tedizolid phosphate. The per protocol statistical approach used in this noncompartmental analysis allowed data collected to generate single concentration listing. As specified in the protocol, AUC0-last for tedizolid metabolite in Part A (Group 1 [Cohorts 1 and 2], Group 2 Cohort 1, Group 2 Cohort 2, Group 3 Cohort 1, Group 3 Cohort 2) were not included in this endpoint and have been reported separately in the record.
Time Frame: 1, 3, 5, 8, 12, and 24 hours post start of dosing
Population: The subset of participants who complied with the protocol to ensure that data exhibits treatment effects, according to the scientific model and had data available for this outcome. AUC0-last for tedizolid metabolite in Part A (Group 1 [Cohorts 1 and 2], Group 2 Cohort 1, Group 2 Cohort 2, Group 3 Cohort 1, Group 3 Cohort 2) are excluded and have been reported separately.
Measure: Number; unit: hr*μg/mL
Arm/Group | Group 1 Cohorts 1+2:SD IV Tedizolid Phosphate 28days-<24months | Part A Group 2 Cohort 1: Single Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 2 Cohort 2: Multiple Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 3 Cohort 1: Single Dose IV Tedizolid Phosphate (Preterm) Birth to <28 Days | Part A Group 3 Cohort 2: Multiple Dose IV Tedizolid Phosphate IV (Preterm) Birth to <28 Days | Part B Group 4: Single Dose Oral Tedizolid Phosphate 28 Days to <24 Months | Part B Group 5: Single Dose Oral Tedizolid Phosphate (Full Term) Birth to <28 Days | Part B Group 6: Single Dose Oral Tedizolid Phosphate (Preterm) Birth to <28 Days
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 3
hr*μg/mL |  |  |  |  |  | 7.92 | 9.25 | 14.9

22. Primary Outcome: Part B: AUC0-inf of Tedizolid (Active Metabolite) After Single-dose Administration of Tedizolid Phosphate Oral Suspension
Description: AUC0-inf of tedizolid (metabolite) was quantified in participants receiving tedizolid phosphate. The per protocol statistical approach used in this noncompartmental analysis allowed data collected to generate single concentration listing. As specified in the protocol, AUC0-inf for tedizolid metabolite in Part A (Group 1 [Cohorts 1 and 2], Group 2 Cohort 1, Group 2 Cohort 2, Group 3 Cohort 1, Group 3 Cohort 2) were not included in this endpoint and have been reported separately in the record.
Time Frame: 1, 3, 5, 8, 12, and 24 hours post start of dosing
Population: The subset of participants who complied with the protocol to ensure that data exhibits treatment effects, according to the scientific model and had data available for this outcome. AUC0-inf for tedizolid metabolite in Part A (Group 1 [Cohorts 1 and 2], Group 2 Cohort 1, Group 2 Cohort 2, Group 3 Cohort 1, Group 3 Cohort 2) are excluded and have been reported separately.
Measure: Number; unit: hr*μg/mL
Arm/Group | Group 1 Cohorts 1+2:SD IV Tedizolid Phosphate 28days-<24months | Part A Group 2 Cohort 1: Single Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 2 Cohort 2: Multiple Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 3 Cohort 1: Single Dose IV Tedizolid Phosphate (Preterm) Birth to <28 Days | Part A Group 3 Cohort 2: Multiple Dose IV Tedizolid Phosphate IV (Preterm) Birth to <28 Days | Part B Group 4: Single Dose Oral Tedizolid Phosphate 28 Days to <24 Months | Part B Group 5: Single Dose Oral Tedizolid Phosphate (Full Term) Birth to <28 Days | Part B Group 6: Single Dose Oral Tedizolid Phosphate (Preterm) Birth to <28 Days
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 3
hr*μg/mL |  |  |  |  |  | 8.36 | 9.44 | 22.1

23. Primary Outcome: Part B: Cmax of Tedizolid (Active Metabolite) After Single-dose Administration of Tedizolid Phosphate Oral Suspension
Description: Cmax of tedizolid (metabolite) was quantified in participants receiving tedizolid phosphate. The per protocol statistical approach used in this noncompartmental analysis allowed data collected to generate single concentration listing. As specified in the protocol, Cmax for tedizolid metabolite in Part A (Group 1 [Cohorts 1 and 2], Group 2 Cohort 1, Group 2 Cohort 2, Group 3 Cohort 1, Group 3 Cohort 2) were not included in this endpoint and have been reported separately in the record.
Time Frame: 1, 3, 5, 8, 12, and 24 hours post start of dosing
Population: The subset of participants who complied with the protocol to ensure that data exhibits treatment effects, according to the scientific model and had data available for this outcome. Cmax for tedizolid metabolite in Part A (Group 1 [Cohorts 1 and 2], Group 2 Cohort 1, Group 2 Cohort 2, Group 3 Cohort 1, Group 3 Cohort 2) are excluded and have been reported separately.
Measure: Number; unit: μg/mL
Arm/Group | Group 1 Cohorts 1+2:SD IV Tedizolid Phosphate 28days-<24months | Part A Group 2 Cohort 1: Single Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 2 Cohort 2: Multiple Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 3 Cohort 1: Single Dose IV Tedizolid Phosphate (Preterm) Birth to <28 Days | Part A Group 3 Cohort 2: Multiple Dose IV Tedizolid Phosphate IV (Preterm) Birth to <28 Days | Part B Group 4: Single Dose Oral Tedizolid Phosphate 28 Days to <24 Months | Part B Group 5: Single Dose Oral Tedizolid Phosphate (Full Term) Birth to <28 Days | Part B Group 6: Single Dose Oral Tedizolid Phosphate (Preterm) Birth to <28 Days
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 3
μg/mL |  |  |  |  |  | 1.32 | 0.899 | 1.22

24. Primary Outcome: Part B: Tmax of Tedizolid (Active Metabolite) After Single-dose Administration of Tedizolid Phosphate Oral Suspension
Description: Tmax of tedizolid (metabolite) was quantified in participants receiving tedizolid phosphate. The per protocol statistical approach used in this noncompartmental analysis allowed data collected to generate single listing. As specified in the protocol, Tmax for tedizolid metabolite in Part A (Group 1 [Cohorts 1 and 2], Group 2 Cohort 1, Group 2 Cohort 2, Group 3 Cohort 1, Group 3 Cohort 2) were not included in this endpoint and have been reported separately in the record.
Time Frame: 1, 3, 5, 8, 12, and 24 hours post start of dosing
Population: The subset of participants who complied with the protocol to ensure that data exhibits treatment effects, according to the scientific model and had data available for this outcome. Tmax for tedizolid metabolite in Part A (Group 1 [Cohorts 1 and 2], Group 2 Cohort 1, Group 2 Cohort 2, Group 3 Cohort 1, Group 3 Cohort 2) are excluded and have been reported separately.
Measure: Number; unit: hr
Arm/Group | Group 1 Cohorts 1+2:SD IV Tedizolid Phosphate 28days-<24months | Part A Group 2 Cohort 1: Single Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 2 Cohort 2: Multiple Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 3 Cohort 1: Single Dose IV Tedizolid Phosphate (Preterm) Birth to <28 Days | Part A Group 3 Cohort 2: Multiple Dose IV Tedizolid Phosphate IV (Preterm) Birth to <28 Days | Part B Group 4: Single Dose Oral Tedizolid Phosphate 28 Days to <24 Months | Part B Group 5: Single Dose Oral Tedizolid Phosphate (Full Term) Birth to <28 Days | Part B Group 6: Single Dose Oral Tedizolid Phosphate (Preterm) Birth to <28 Days
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 3
hr |  |  |  |  |  | 1 | 3.03 | 8

25. Primary Outcome: Part B: t½ of Tedizolid (Active Metabolite) After Single-dose Administration of Tedizolid Phosphate Oral Suspension
Description: t½ of tedizolid (metabolite) was quantified in participants receiving tedizolid phosphate. The per protocol statistical approach used in this noncompartmental analysis allowed data collected to generate single listing. As specified in the protocol, t½ for tedizolid metabolite in Part A (Group 1 [Cohorts 1 and 2], Group 2 Cohort 1, Group 2 Cohort 2, Group 3 Cohort 1, Group 3 Cohort 2) were not included in this endpoint and have been reported separately in the record.
Time Frame: 1, 3, 5, 8, 12, and 24 hours post start of dosing
Population: The subset of participants who complied with the protocol to ensure that data exhibits treatment effects, according to the scientific model and had data available for this outcome. t1/2 for tedizolid metabolite in Part A (Group 1 [Cohorts 1 and 2], Group 2 Cohort 1, Group 2 Cohort 2, Group 3 Cohort 1, Group 3 Cohort 2) are excluded and have been reported separately.
Measure: Number; unit: hr
Arm/Group | Group 1 Cohorts 1+2:SD IV Tedizolid Phosphate 28days-<24months | Part A Group 2 Cohort 1: Single Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 2 Cohort 2: Multiple Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 3 Cohort 1: Single Dose IV Tedizolid Phosphate (Preterm) Birth to <28 Days | Part A Group 3 Cohort 2: Multiple Dose IV Tedizolid Phosphate IV (Preterm) Birth to <28 Days | Part B Group 4: Single Dose Oral Tedizolid Phosphate 28 Days to <24 Months | Part B Group 5: Single Dose Oral Tedizolid Phosphate (Full Term) Birth to <28 Days | Part B Group 6: Single Dose Oral Tedizolid Phosphate (Preterm) Birth to <28 Days
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 3
hr |  |  |  |  |  | 5.73 | 3.82 | 13.4

26. Secondary Outcome: Number of Participants With an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants experiencing an AE was reported for each arm.
Time Frame: Up to approximately 21 days
Population: All participants who received at least one dose of the investigational drug were assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A Group 1 Cohort 1: Single Dose IV Tedizolid Phosphate 28 Days to <6 Months | Part A Group 1 Cohort 2: Single Dose IV Tedizolid Phosphate 6 Months to <24 Months | Part A Group 2 Cohort 1: Single Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 2 Cohort 2: Multiple Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 3 Cohort 1: Single Dose IV Tedizolid Phosphate (Preterm) Birth to <28 Days | Part A Group 3 Cohort 2: Multiple Dose IV Tedizolid Phosphate IV (Preterm) Birth to <28 Days | Part B Group 4: Single Dose Oral Tedizolid Phosphate 28 Days to <24 Months | Part B Group 5: Single Dose Oral Tedizolid Phosphate (Full Term) Birth to <28 Days | Part B Group 6: Single Dose Oral Tedizolid Phosphate (Preterm) Birth to <28 Days
Number analyzed (Participants) | 4 | 6 | 8 | 4 | 9 | 4 | 4 | 4 | 4
Participants | 1 | 1 | 0 | 0 | 2 | 2 | 1 | 0 | 1

27. Secondary Outcome: Number of Participants That Discontinued Study Treatment Due to an AE
Description: An AE was defined as any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants that discontinued study treatment due to an AE was reported for each arm.
Time Frame: Up to approximately 3 days
Population: All participants who received at least one dose of the investigational drug were assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A Group 1 Cohort 1: Single Dose IV Tedizolid Phosphate 28 Days to <6 Months | Part A Group 1 Cohort 2: Single Dose IV Tedizolid Phosphate 6 Months to <24 Months | Part A Group 2 Cohort 1: Single Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 2 Cohort 2: Multiple Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 3 Cohort 1: Single Dose IV Tedizolid Phosphate (Preterm) Birth to <28 Days | Part A Group 3 Cohort 2: Multiple Dose IV Tedizolid Phosphate IV (Preterm) Birth to <28 Days | Part B Group 4: Single Dose Oral Tedizolid Phosphate 28 Days to <24 Months | Part B Group 5: Single Dose Oral Tedizolid Phosphate (Full Term) Birth to <28 Days | Part B Group 6: Single Dose Oral Tedizolid Phosphate (Preterm) Birth to <28 Days
Number analyzed (Participants) | 4 | 6 | 8 | 4 | 9 | 4 | 4 | 4 | 4
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to approximately 21 days
Description: Safety: All participants who received at least one dose of the investigational drug.
  All-cause mortality: All allocated participants.
Arm/Group | Part A Group 1 Cohort 1: Single Dose IV Tedizolid Phosphate 28 Days to <6 Months | Part A Group 1 Cohort 2: Single Dose IV Tedizolid Phosphate 6 Months to <24 Months | Part A Group 2 Cohort 1: Single Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 2 Cohort 2: Multiple Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days | Part A Group 3 Cohort 1: Single Dose IV Tedizolid Phosphate (Preterm) Birth to <28 Days | Part A Group 3 Cohort 2: Multiple Dose IV Tedizolid Phosphate IV (Preterm) Birth to <28 Days | Part B Group 4: Single Dose Oral Tedizolid Phosphate 28 Days to <24 Months | Part B Group 5: Single Dose Oral Tedizolid Phosphate (Full Term) Birth to <28 Days | Part B Group 6: Single Dose Oral Tedizolid Phosphate (Preterm) Birth to <28 Days
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/6 | 0/8 | 0/4 | 0/9 | 0/4 | 0/4 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/6 | 0/8 | 0/4 | 0/9 | 0/4 | 0/4 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 1/6 | 0/8 | 0/4 | 2/9 | 2/4 | 1/4 | 0/4 | 1/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A Group 1 Cohort 1: Single Dose IV Tedizolid Phosphate 28 Days to <6 Months (N=4) | Part A Group 1 Cohort 2: Single Dose IV Tedizolid Phosphate 6 Months to <24 Months (N=6) | Part A Group 2 Cohort 1: Single Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days (N=8) | Part A Group 2 Cohort 2: Multiple Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days (N=4) | Part A Group 3 Cohort 1: Single Dose IV Tedizolid Phosphate (Preterm) Birth to <28 Days (N=9) | Part A Group 3 Cohort 2: Multiple Dose IV Tedizolid Phosphate IV (Preterm) Birth to <28 Days (N=4) | Part B Group 4: Single Dose Oral Tedizolid Phosphate 28 Days to <24 Months (N=4) | Part B Group 5: Single Dose Oral Tedizolid Phosphate (Full Term) Birth to <28 Days (N=4) | Part B Group 6: Single Dose Oral Tedizolid Phosphate (Preterm) Birth to <28 Days (N=4)
Therapeutic product effect incomplete (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A Group 1 Cohort 1: Single Dose IV Tedizolid Phosphate 28 Days to <6 Months (N=4) | Part A Group 1 Cohort 2: Single Dose IV Tedizolid Phosphate 6 Months to <24 Months (N=6) | Part A Group 2 Cohort 1: Single Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days (N=8) | Part A Group 2 Cohort 2: Multiple Dose IV Tedizolid Phosphate (Full Term) Birth to <28 Days (N=4) | Part A Group 3 Cohort 1: Single Dose IV Tedizolid Phosphate (Preterm) Birth to <28 Days (N=9) | Part A Group 3 Cohort 2: Multiple Dose IV Tedizolid Phosphate IV (Preterm) Birth to <28 Days (N=4) | Part B Group 4: Single Dose Oral Tedizolid Phosphate 28 Days to <24 Months (N=4) | Part B Group 5: Single Dose Oral Tedizolid Phosphate (Full Term) Birth to <28 Days (N=4) | Part B Group 6: Single Dose Oral Tedizolid Phosphate (Preterm) Birth to <28 Days (N=4)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Swelling of eyelid (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Serratia sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Immature granulocyte count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-06): https://cdn.clinicaltrials.gov/large-docs/65/NCT03217565/Prot_SAP_000.pdf